CLINICAL TRIAL: NCT01136772
Title: A Comparison of Long-Acting Injectable Medications for Schizophrenia
Acronym: ACLAIMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Duke University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #6017; R01MH081107 (NIH)
Record Dates: First submitted 2010-05-14; First posted 2010-06-03 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — haloperidol decanoate; Haloperidol; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paliperidone palmitate (Experimental): Intramuscular injections of paliperidone palmitate 39-234 mg every month
  Interventions: Drug: paliperidone palmitate
- Haloperidol decanoate (Active Comparator): Intramuscular injections of haloperidol decanoate 25-200 mg every month
  Interventions: Drug: haloperidol decanoate

INTERVENTIONS:
Drug: haloperidol decanoate — haloperidol decanoate injections, 25-200 mg once a month
  Other Names: Haldol
  Arms: Haloperidol decanoate
Drug: paliperidone palmitate — Paliperidone palmitate injections, 39 mg - 234 mg once a month
  Other Names: Invega Sustenna
  Arms: Paliperidone palmitate

SUMMARY:
The purpose of this research study is to compare the "real-world" effectiveness of two FDA-approved and widely used long-acting injectable antipsychotic medications (paliperidone palmitate and haloperidol decanoate) in patients with schizophrenia or schizoaffective disorder who are expected to benefit from the improved medication compliance associated with injectable medications. The goal is to evaluate the effects of the medications on outcomes of importance to patients (relapse, symptoms, adverse effects, functioning) as well as policy makers (all of the above plus costs).

DETAILED DESCRIPTION:
The purpose of this comparative effectiveness research study is to learn more about different medications called antipsychotics that are used to treat schizophrenia or schizoaffective disorder. Specifically, we are looking at long-acting medications that are given by injection every month, instead of being taken by mouth every day. In this multi-site study, we are comparing the risk and benefits of two FDA-approved long-acting injectable medications (paliperidone palmitate and haloperidol decanoate). Study participants with schizophrenia or schizoaffective disorder are expected to benefit from the improved medication schedule.

This study aims to enroll 360 individuals with schizophrenia or schizoaffective disorder for whom treatment with a long-acting injectable antipsychotic medication is likely to be helpful. Study participants will be randomly assigned to treatment with either paliperidone palmitate and haloperidol decanoate for up to 24 months. Participants will have an equal chance of being assigned to each medication, however participants will not know which medication they are taking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder as defined by DSM-IV-TR criteria
* Age 18-65 years
* Capacity to provide informed consent
* Patients who are likely to benefit from treatment with long-acting injectable paliperidone palmitate or haloperidol decanoate
* Women of child bearing potential must have a negative serum pregnancy test at the Screening Visit.

Exclusion Criteria:

* Patients who are currently stable and doing well on an antipsychotic regimen
* Patients not expected to benefit from the study medications due to past experience with risperidone, paliperidone or haloperidol
* Patients with tardive dyskinesia that is moderate or severe
* Patients with any medical condition that, in the judgment of the investigator, might preclude safe completion of the study
* Women who are pregnant or breastfeeding
* Patients with mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Stroup, MD, MPH, Principal Investigator — Columbia University; Joseph P McEvoy, MD, Principal Investigator — Duke University
Locations (22):
- United States (22):
  - VA Palo Alto Heathcare Systems, Palo Alto, California
  - Yale University/Connecticut Mental Health Center, New Haven, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - University of Iowa Hospital, Iowa City, Iowa
  - Clinical Research Institute, Wichita, Kansas
  - Clinical Insights, Inc., Glen Burnie, Maryland
  - John D. Dingell VA Medical Center, Detroit, Michigan
  - Sparrow St. Lawrence Hospital, Michigan State University Psychiatry, Lansing, Michigan
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Creighton University Dept. of Psychiatry, Omaha, Nebraska
  - Research Foundation for Mental Hygiene, New York, New York
  - University of Rochester, Rochester, New York
  - John Umstead Hospital/Duke University, Butner, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Behavioral Care, Durham, North Carolina
  - Louis Stokes Cleveland VA Medical Center, Brecksville, Ohio
  - Philadelphia VA Medical Center-116A, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Central Texas Veterans Health Care System, Waco, Texas
  - Frontier Institute, Spokane, Washington
  - VA Puget Sound Health Care System, Tacoma, Washington

REFERENCES:
- [Result] McEvoy JP, Byerly M, Hamer RM, Dominik R, Swartz MS, Rosenheck RA, Ray N, Lamberti JS, Buckley PF, Wilkins TM, Stroup TS. Effectiveness of paliperidone palmitate vs haloperidol decanoate for maintenance treatment of schizophrenia: a randomized clinical trial. JAMA. 2014 May 21;311(19):1978-87. doi: 10.1001/jama.2014.4310. PMID 24846035
- [Result] Rosenheck RA, Leslie DL, Sint KJ, Lin H, Li Y, McEvoy JP, Byerly MJ, Hamer RM, Swartz MS, Stroup TS. Cost-Effectiveness of Long-Acting Injectable Paliperidone Palmitate Versus Haloperidol Decanoate in Maintenance Treatment of Schizophrenia. Psychiatr Serv. 2016 Oct 1;67(10):1124-1130. doi: 10.1176/appi.ps.201500447. Epub 2016 Jun 1. PMID 27247177
- [Derived] Stroup TS, Bareis NA, Rosenheck RA, Swartz MS, McEvoy JP. Heterogeneity of Treatment Effects of Long-Acting Injectable Antipsychotic Medications. J Clin Psychiatry. 2018 Nov 27;80(1):18m12109. doi: 10.4088/JCP.18m12109. PMID 30549494

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paliperidone Palmitate | Haloperidol Decanoate
Started | 157 | 154
Safety Population | 147 (Includes all randomized participants who received at least one dose of the injectable medication) | 147 (Includes all randomized participants who received at least one dose of the injectable medication)
Completed | 41 | 44
Not Completed | 116 | 110
Not completed — Adverse Event | 15 | 14
Not completed — Lack of Efficacy | 42 | 39
Not completed — Administrative | 14 | 12
Not completed — Withdrawal by Subject | 33 | 36
Not completed — Did not receive injection | 10 | 7
Not completed — Did not follow up after first injection | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of modified intent-to-treat population (those who received at least one injection and attended one follow-up appointment)
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone Palmitate | Haloperidol Decanoate | Total
Number analyzed (Participants) | 145 | 145 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (12.6) | 45 (12.3) | 44 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 106 | 110 | 216

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Failure
Description: Efficacy failure as indicated by psychiatric hospitalization, need for crisis intervention, clinical decision that oral antipsychotic medication cannot be discontinued in less than eight weeks, a clinical decision to discontinue the medication due to inadequate benefit, or the ongoing or repeated need for adjunctive antipsychotic medication.
Time Frame: 24 months
Population: All randomized participants who received an injection and attended one follow-up appointment
Measure: Number; unit: participants
Arm/Group | Paliperidone Palmitate | Haloperidol Decanoate
Number analyzed (Participants) | 145 | 145
participants | 49 | 47

2. Secondary Outcome: Changes in Psychiatric Symptoms
Description: The Positive and Negative Syndrome Scale measures the core symptoms associated with schizophrenia. The measure includes 30 items rated from 1=absent to 7=extremely severe. Full range of scores is 30-210 with higher scores representing more severe illness. Reductions in symptoms over time represent improvement.
Time Frame: Baseline to 6 months
Population: Participants with PANSS scores at 6 months
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Haloperidol Decanoate
Number analyzed (Participants) | 91 | 88
Units on a scale | -6.87 [-8.79 to -4.94] | -6.40 [-8.32 to -4.48]

ADVERSE EVENTS:
Arm/Group | Paliperidone Palmitate | Haloperidol Decanoate
Serious Adverse Events (participants affected / at risk) | 53/147 | 45/147
Other Adverse Events (participants affected / at risk) | 100/147 | 88/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=147) | Haloperidol Decanoate (N=147)
Suicidal ideation (Psychiatric disorders) | 20 | 16
Suicidal Act (Psychiatric disorders) | 2 | 5
Homicidal ideation (Psychiatric disorders) | 8 | 7
Homocidal Act (Psychiatric disorders) | 0 | 1
Violent ideation (Psychiatric disorders) | 2 | 3
Violent act (Psychiatric disorders) | 0 | 2
Psychiatric hospitalization (Psychiatric disorders) | 44 | 34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=147) | Haloperidol Decanoate (N=147)
Insomnia (Psychiatric disorders) | 49 | 54 — Events rated moderate or severe
Sleepiness (Psychiatric disorders) | 41 | 44 — Events rated moderate or severe
Dry mouth (Gastrointestinal disorders) | 40 | 34 — Events rated moderate or severe
Increased appetite (General disorders) | 33 | 26 — Events rated moderate or severe
Hypersomnia (Psychiatric disorders) | 24 | 20 — Events rated moderate or severe
Sialorrhea (General disorders) | 24 | 16 — Events rated moderate or severe
Constipation (Gastrointestinal disorders) | 21 | 20 — Events rated moderate or severe
Orthostatic faintness (Cardiac disorders) | 14 | 12 — Events rated moderate or severe
Incontinence/nocturia (Renal and urinary disorders) | 13 | 8 — Events rated moderate or severe
Menstrual irregularities (Reproductive system and breast disorders) | 12 | 5 — Events rated moderate or severe
Urinary hesitancy (Renal and urinary disorders) | 7 | 9 — Events rated moderate or severe

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No